CLINICAL TRIAL: NCT02936141
Title: Psychosocial Intervention Targeting Homeless With Mental Disorders in the City of Maputo and Matola: a Study Protocol
Brief Title: Psychosocial Intervention Designed to Familial Reintegration of Homeless With Mental Disorder in Maputo and Matola City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Mozambique (Other Government)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DSM-000-RS
Record Dates: First submitted 2016-09-27; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Mental Disorders
Keywords: homeless, mental disorders, attendance
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy, Group; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group psychotherapy (Experimental): Group psychotherapy sessions includes the following: training of social skills (such as communication, social interaction and assertive behaviors), cognitive stimulation and training of activities of daily living (such as personal hygiene, hygiene of spaces and standardized mealtimes)
  Interventions: Behavioral: Group psychotherapy

INTERVENTIONS:
Behavioral: Group psychotherapy — Includes a group (up to 10 participants) weekly session with a duration of 90 minutes where it is stimulated communication, adaptative behaviour and social living
  Other Names: Cognitive Therapy

SUMMARY:
The aim of this project is to describe the mental health status of the homeless people in Maputo and Matola utilising standardised clinical and socio-demographic assessments. Simultaneously; the study aims to determine the influence of a psychosocial intervention in patients with apparent signs of mental illness, aiming at his/her family reintegration; This study is conducted hypothesizing that the familial reintegration after intervention would be the same across patients with different mental disorders.

DETAILED DESCRIPTION:
Even though the Mental Health Program in Mozambique have been providing and implementing services to reduce the gap in the treatment of mental disorders, there are no specific programs for homeless people. Additionally, in the country, there are no specific interventions for the homeless mentally ill, combining hospital and community interventions. Therefore we designed a pilot study to evaluate the profile of those individuals who live on the streets with apparent mental illness, and the effectiveness of the intervention plan considered for this purpose. Utilising an intervention study in community and hospital settings, we aim to understand the mental health status of the homeless people and appraise the effectiveness and acceptability of a multidisciplinary intervention in a low-income country. Our main hypothesis is that the intervention designed to facilitate and maintain the homeless people with mental health disorders in treatment through the implementation of evidence-based intervention can increase the reintegration of homeless people in their community, and that the familial reintegration would be the same among patients with different mental disorders. The present study was waived of approval by the National Bioethics Committee for Health, since it was realized on behalf of an activity held by the Ministry of Health. The study will be conducted in Maputo and Matola cities both in the southern region of Mozambique. These cities were chosen because of their accessibility and due to the dimension of the homeless population, representing an urban and suburban area respectively. The selection of the sample of homeless will be by convenience. After a period of mapping (to study homeless' routines including usual pathways), potential participants and their relatives will be approached. Members of the community such as the head of the block and member of the neighborhood will be involved to facilitate the family contact that after explanation about the goals of the program will be asked to give their consent; later the potential participant will be approached on the street and informed about the objectives of the program, the length of the study, any benefits or risk they might incur as participants, who to contact in case they have questions or concerns and their right to decline to participate without coercion. Then, they will be proposed referral to inpatient unit where it will be done the psychological and medical treatment, rehabilitation and family reintegration and will be asked to give their informed consent as well. Upon arrival to the psychiatric hospital, a multidisciplinary assistance team will welcome the homeless by initiating the intervention with the personal hygiene, including shave and haircut. The diagnosis will be established by experienced psychiatrists, using a structured diagnostic assessment instrument - Mini International Neuropsychiatric Interview (MINI) - and a socio-demographic inventory (with data such as age, name, gender, marital status, occupation, education, employment, religion and economic conditions). After psychiatric evaluation, participants will initiate psychopharmacological treatment according to the needs of each patient. Laboratorial analyses will be performed to exclude organic diseases, and in positive cases an additional clinical examination will be requested. Once the symptoms are controlled, the patients will be submitted to a psychological evaluation and initiate group psychotherapy interventions. Group psychotherapy sessions included the following: training of social skills (such as communication, social interaction and assertive behaviors); cognitive stimulation and training of activities of daily living (such as personal hygiene, hygiene of spaces and standardized mealtimes). In a subsequent phase, for the family reintegration preparation process, group psychotherapy sessions and psychoeducation will be held involving patients' relatives.

Furthermore social workers in coordination with the community leaders and the municipal authorities will ask for permission to do home visits to the relatives of the participants so as to create the appropriated environment to the family reintegration process. Throughout these visits, the level of family involvement regarding the therapeutic process, the patient's health status, and the search information of their family member's disease will be assessed. Family reintegration refers to the process of return from an institution or shelter to the original, extensive or adopted family. In our study, we consider family reintegration as the return of the participant to family of origin after completing the intervention at the hospital level.

After the family reintegration it will be made a follow up every 3 months during 12 months. Participants will be registered and followed in clinic in nearby sanitary units of their residence areas as usual procedure after discharge of patients of the psychiatric unity.

Data analysis will be performed using the Statistical Package for Social Sciences version 22, for the quantitative data analysis. All the collected information will be coded including the identification of patients, relatives, health professionals and community leaders involved in the study.

ELIGIBILITY:
Inclusion Criteria:

- People with apparent signs of mental disorder, who had been living on the street for more than 30 days who agreed to sign or give a verbal consent (by herself/himself, family/relatives)

Exclusion Criteria:

* Homeless persons without apparent signs of mental illness, with obvious physical illness, seemingly under the age of 18 and that were not able to give informed consent/those who it was not possible to contact their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Familial reintegration | Every three months after discharge during 12 months
  The return of the participant to family of origin after completing the intervention at the hospital level. This outcome was based on the questionnaire: "inquiry homeless data collection", drawn for the study. It contains a dichotomized question: patient living with the relatives during the first visit (yes or no), second visit (yes or no) and third visit (yes or no) throughout follow-up visits. When the answer was yes in three consecutive visits, he/she was considered reintegrated in the family in the present study.

SECONDARY OUTCOMES:
Social skills | Every three months after discharge during 12 months
  Components of social skills were accessed through adaptation of Social Skills Evaluation Scales (EEHS - Tremblay & Bandeira, 1989) to the mozambican cultural context. The items considered included: verbal skills, conflict resolution and non-verbal skills. This evaluation was made in the beginning of treatment and during the follow-up home visits by trained social workers and psychologists.

CONTACTS AND LOCATIONS:
Overall Officials: Lídia C. Gouveia, MD, Principal Investigator — Mental Health Department of Ministry of Health

IPD SHARING:
Plan to Share IPD: Yes
There is a need of reformulating database so as to better protect participant's confidentiality

REFERENCES:
- [Background] Patel V, Simbine AP, Soares IC, Weiss HA, Wheeler E. Prevalence of severe mental and neurological disorders in Mozambique: a population-based survey. Lancet. 2007 Sep 22;370(9592):1055-60. doi: 10.1016/S0140-6736(07)61479-2. PMID 17889244
- [Result] Patra S, Anand K. Homelessness: a hidden public health problem. Indian J Public Health. 2008 Jul-Sep;52(3):164-70. PMID 19189843
- [Result] Dennis DL, Buckner JC, Lipton FR, Levine IS. A decade of research and services for homeless mentally ill persons. Where do we stand? Am Psychol. 1991 Nov;46(11):1129-38. doi: 10.1037//0003-066x.46.11.1129. PMID 1772150
- [Result] Scott J. Homelessness and mental illness. Br J Psychiatry. 1993 Mar;162:314-24. doi: 10.1192/bjp.162.3.314. PMID 8453425
- [Result] Sullivan G, Burnam A, Koegel P. Pathways to homelessness among the mentally ill. Soc Psychiatry Psychiatr Epidemiol. 2000 Oct;35(10):444-50. doi: 10.1007/s001270050262. PMID 11127718
- [Result] Folsom DP, Hawthorne W, Lindamer L, Gilmer T, Bailey A, Golshan S, Garcia P, Unutzer J, Hough R, Jeste DV. Prevalence and risk factors for homelessness and utilization of mental health services among 10,340 patients with serious mental illness in a large public mental health system. Am J Psychiatry. 2005 Feb;162(2):370-6. doi: 10.1176/appi.ajp.162.2.370. PMID 15677603